CLINICAL TRIAL: NCT01757522
Title: Detection of Right Ventricular Dysfunction by 2D Strain During Acute Respiratory Distress Syndrom (ARDS)
Acronym: STRAIN
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-A01204-39
Record Dates: First submitted 2012-12-04; First posted 2012-12-31 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-05

CONDITIONS: Acute Respiratory Distress Syndrome; Right Ventricular Dysfunction; Right Heart Failure; Acute Cor Pulmonale
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventricular Dysfunction, Right; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasmatic levels of NT proBNP and pre pro endothelin are monitored in ARDS group to determine whether these biomarkers can help detect right ventricular dysfunction.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ARDS group: Patients under mechanical ventilation since less than 24 hours at inclusion and presenting acute respiratory distress syndrome criteria.
- ALI group: Patients under mechanical ventilation and presenting acute lung injury criteria.
- Control Group: Patients under mechanical ventilation for a non-respiratory cause

SUMMARY:
Acute respiratory distress syndrome (ARDS) and mechanical ventilation can lead to right ventricular dysfunction and ultimately right ventricular failure by increasing pulmonary vascular resistances and pressure load. This can be prevented by modifying ventilator settings, using vasopressors or inotropes or even by prone positionning.But to do so, right ventricular dysfonction has to be detected. Echocardiography has emerged as a first line tool to diagnose right heart failure. Recently, strain analysis showed promising results to detect early right ventricle abnormalities in other settings such as pulmonary hypertension or scleroderma. We therefore decided to determine whether 2D strain could help detect early right ventricular dysfunction in ARDS.

ELIGIBILITY:
ARDS group

Inclusion Criteria:

* Need for mechanical ventilation
* ARDS criteria met: Respiratory failure not fully explained by cardiac failure, Pao2/FiO2<200, bilateral opacities on Chest imaging, all symptoms appeared within 1 week

Exclusion Criteria:

* Predictable duration of mechanical ventilation shorter than 48 hours
* Contraindication to transesophageal echocardiography

ALI group:

Inclusion Criteria:

* Need for mechanical ventilation
* ALI criteria met: Respiratory failure not fully explained by cardiac failure, Pao2/FiO2<300, bilateral opacities on Chest imaging, all symptoms appeared within 1 week

Exclusion Criteria:

* Predictable duration of mechanical ventilation shorter than 48 hours

Control Group:

Inclusion Criteria:

* Need for mechanical ventilation for a non-respiratory cause

Exclusion Criteria:

* Need for FiO2>30%
* Known cardiac abnormalities
* Cardiac drugs intake during last 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited in our medical intensive care unit at Grenoble University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2013-01-03 (Actual); Primary Completion 2015-03-17 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Right ventricle 2D strain | Duration of mechanical ventilation
  We will assess whether 2D strain can detect a right ventricular dysfunction as compared to standard echocardiographic parameters

SECONDARY OUTCOMES:
Mean right ventricle strain under ventilated patients | at inclusion
  We measure right ventricle strain (RV strain) in patients under mechanical ventilation for a non-respiratory cause. This allows us to determine the mean value of RV strain under ventilation when there is no respiratory failure.
Reproducibility between transthoracic and transesophageal strain measures | Time of mechanical ventilation
  In ARDS patients, we record a transthoracic and transesophageal echocardiography. We compare RV strain values obtained from transthoracic and transesophageal echocardiography.
NT pro BNP and pre pro endothelin plasma level | At inclusion in ARDS patients
  These assays are made based on the hypothesis they could help discriminate between patients who will develop a right ventricular dysfunction from those who will not. A blood sample is withdrawn at the same time as echocardiography only in the ARDS group.

CONTACTS AND LOCATIONS:
Overall Officials: Carole SCHWEBEL, PU/PH, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital of Grenoble, Grenoble, Cedex 09, France